CLINICAL TRIAL: NCT02325154
Title: Cerebral Near-Infrared Spectroscopy and Hypotensive Anesthesia in Patients Undergoing Total Hip Arthroplasty
Brief Title: Cerebral Oxygenation in Total Hip Arthroplasty Patients
Acronym: THANIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-047
Record Dates: First submitted 2014-12-04; First posted 2014-12-24 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Oxygen Desaturation; Post-operative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- THA Patients (Experimental): Patients undergoing unilateral total hip arthroplasty
  Interventions: Device: Cerebral Oximeter

INTERVENTIONS:
Device: Cerebral Oximeter — Use of cerebral oximeter to monitor cerebral oxygenation for occurence of desaturation events.
  Other Names: oximeter

SUMMARY:
We plan to investigate the relationship between hypotensive epidural anesthesia for hip arthroplasty and cerebral oxygen saturation.

DETAILED DESCRIPTION:
The relationship between cerebral oxygenation and blood pressure in patients undergoing hypotensive epidural anesthesia has not been completely elucidated. Previous publications have demonstrated a low incidence of post-op cognitive dysfunction in patients undergoing hypotensive epidural anesthesia for total hip replacement (1-3) and that cerebral blood flow velocity is preserved as measured by transcranial Doppler (4). An earlier investigation by Dr. Yadeau demonstrated infrequent cerebral oxygen desaturation in spontaneously breathing patients undergoing shoulder arthroscopy, even in the presence of hypotension (4), but did not investigate outcomes in the cognitive domain or have a control group of patients undergoing surgery with general anesthesia. There has only been one study looking at cerebral oxygenation and hip surgery, which was performed in elderly patients with fractures. It demonstrated that patients with low pre-op regional cerebral oxygen saturation (rSO2) had higher incidence of delirium (5) but many of those patients had surgery under general anesthesia. Given the costs associated with post-op delirium, cognitive dysfunction and stroke (6) and based on the fact that previous publications from this institution have demonstrated both a low incidence of cognitive dysfunction and preservation of cerebral blood flow velocity using this anesthetic technique, we hypothesized that cerebral oxygen desaturation will not occur in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18-80 years old undergoing unilateral total hip arthroplasty
* Hypotensive epidural anesthesia

Exclusion Criteria:

* Contraindication to controlled hypotension and/or neuraxial anesthesia.
* Severe pulmonary hypertension or pre-op systolic blood pressure reading >150 mm Hg
* Moderate to severe valvular stenosis.
* History of stroke, dementia, or post-op delirium
* Prior OSA diagnosis
* History of benzodiazepine use (regular use for longer than 3 months)
* Chronic renal or hepatic disease (renal failure, history of liver failure, cirrhosis)
* History of alcoholism or heavy alcohol intake (defined as averaging more than 3 drinks per night; recovery is OK)
* Parkinson's disease
* Severe chronic pulmonary disease
* Total anterior hip approach being used
* Hip resurfacing procedure
* Non-English Speaking*

  * Questionnaires being used to assess mental status are only validated in English.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sean Garvin, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Williams-Russo P, Sharrock NE, Mattis S, Szatrowski TP, Charlson ME. Cognitive effects after epidural vs general anesthesia in older adults. A randomized trial. JAMA. 1995 Jul 5;274(1):44-50. PMID 7791257
- [Result] Sharrock NE, Fischer G, Goss S, Flynn E, Go G, Sculco TP, Salvati EA. The early recovery of cognitive function after total-hip replacement under hypotensive epidural anesthesia. Reg Anesth Pain Med. 2005 Mar-Apr;30(2):123-7. doi: 10.1016/j.rapm.2004.12.005. PMID 15765453
- [Result] Rade MC, Yadeau JT, Ford C, Reid MC. Postoperative delirium in elderly patients after elective hip or knee arthroplasty performed under regional anesthesia. HSS J. 2011 Jul;7(2):151-6. doi: 10.1007/s11420-011-9195-2. Epub 2011 Feb 11. PMID 22754416
- [Result] Yadeau JT, Liu SS, Bang H, Shaw PM, Wilfred SE, Shetty T, Gordon M. Cerebral oximetry desaturation during shoulder surgery performed in a sitting position under regional anesthesia. Can J Anaesth. 2011 Nov;58(11):986-92. doi: 10.1007/s12630-011-9574-7. Epub 2011 Aug 25. PMID 21866430
- [Result] Papadopoulos G, Karanikolas M, Liarmakopoulou A, Papathanakos G, Korre M, Beris A. Cerebral oximetry and cognitive dysfunction in elderly patients undergoing surgery for hip fractures: a prospective observational study. Open Orthop J. 2012;6:400-5. doi: 10.2174/1874325001206010400. Epub 2012 Sep 3. PMID 22962570
- [Result] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Result] Murphy GS, Szokol JW, Marymont JH, Greenberg SB, Avram MJ, Vender JS, Vaughn J, Nisman M. Cerebral oxygen desaturation events assessed by near-infrared spectroscopy during shoulder arthroscopy in the beach chair and lateral decubitus positions. Anesth Analg. 2010 Aug;111(2):496-505. doi: 10.1213/ANE.0b013e3181e33bd9. Epub 2010 May 27. PMID 20508134

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | THA Patients
Started | 100
Completed | 99
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | THA Patients
Number analyzed (Participants) | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Categories: Black or African American | 4
  Race Categories: White | 86
  Race Categories: Unknown | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Desaturation Incidences
Description: The number of participant's experiencing an intra-operative cerebral oxygen desaturation event.
  Measured in the number of patients, beginning with the time the patients' enters the operating room and up to 4 hours.
Time Frame: Intra-operation (when the patient enters the operating room, up to 4 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | THA Patients
Number analyzed (Participants) | 99
Participants | 4

2. Secondary Outcome: Duration of Oxygen Desaturation
Description: Duration of cerebral oxygen desaturation
Time Frame: Intra-op ( during the time the patient is in the operating room, up to 4 hours)
Population: only 4 patients had desaturation events
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | THA Patients
Number analyzed (Participants) | 4
seconds | 11 [5 to 120]

3. Secondary Outcome: Presence of Post-operative Delirium
Description: The number of patients who have post-operative delirium, as determined by counting the patients who suffer from this condition.
  Although recorded at various time points, the total number of participants experiencing post-operative delirium was summed and reported.
Time Frame: Post-op Day 1, Post-op Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | THA Patients
Number analyzed (Participants) | 99
Participants | 0

4. Secondary Outcome: Patients With Cognitive Dysfunction
Description: The number of patients considered to experience cognitive dysfunction as identified by low scores on the mini-Cog.
  The Mini-Cog checks for the brain function (or the cognitive impairment) of the participant. The Mini-Cog does this by examining a patient's ability in two areas. This is done via a three-word recall test and the Clock Drawing Test.
  1. Three-Word Recall
  2. The Clock Drawing Test (CDT)
  There are five total points a person can score on the Mini-Cog:
  * Give one point for each word that was correctly remembered. (0-3 points)
  * Give two points for a correctly drawn clock, meaning the numbers are in roughly the correct locations and two hands are pointed to the 11 and the 2. The length of the hands does not matter. (0 or 2 points) If a patient scores less than three points, they are counted as experiencing cognitive dysfunction.
  Although collected across different time points, the total number of patients scoring less than 3 points were summed and reported.
Time Frame: Post-op Day 1, Post-op Day 2
Population: From baseline to POD 1, 7 patients had positive scores in Mini-Cog Test. On POD 2, one patient withdrew from the study, so 6 patients reported positive scores in Mini-Cog test.
Measure: Count of Participants; unit: Participants
Arm/Group | THA Patients
Number analyzed (Participants) | 99
Participants
  Post-Operative Day 1: number analyzed (Participants) | 7
  Post-Operative Day 1: Abnormal Clock Drawing From baseline | 3
  Post-Operative Day 1: Word Recall decrease From baseline | 4
  Post-Operative Day 2: number analyzed (Participants) | 6
  Post-Operative Day 2: Abnormal Clock Drawing From baseline | 3
  Post-Operative Day 2: Word Recall decrease From baseline | 3

ADVERSE EVENTS:
Time Frame: up to 2 days following surgery
Arm/Group | THA Patients
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes